CLINICAL TRIAL: NCT05623917
Title: Sleep Quality, Stress/Depression, Autonomic Responses to Breathing Exercise in Systemic Sclerosis
Brief Title: Sleep Quality, Stress, Depression, Blood Pressure Responses to Diaphragmatic Respiratory Exercise in Systemic Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004115
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercised group (Experimental): the group will contain 20 females. the females will receive tele-supervised Diaphragmatic Respiratory Exercise ( applied at the homes of the females two times per the day, at the morning and at the evening, twenty minutes for every time, the sessions will be applied daily for 3 months in all females).
  Interventions: Behavioral: Tele-supervised diaphragmatic respiratory exercise
- control group (No Intervention): he females in the this group will be waiting-list control females who will receive no training.

INTERVENTIONS:
Behavioral: Tele-supervised diaphragmatic respiratory exercise — the group will contain 20 females. the females will receive tele-supervised Diaphragmatic Respiratory Exercise ( applied at the homes of the females two times per the day, at the morning and at the evening, twenty minutes for every time, the sessions will be applied daily for 3 months in all females).
  Arms: Exercised group

SUMMARY:
systemic sclerosis women usually report problems such as stress/depression, fatigue, not deep sleep. complementary therapies may improve the reported problems in those patients

DETAILED DESCRIPTION:
the assignment of females with systemic sclerosis (n= forty females) to two equal groups. the group will contain 20 females. the first group will receive tele-supervised Diaphragmatic Respiratory Exercise ( applied at the homes of the females two times per the day, at the morning and at the evening, twenty minutes for every time, the sessions will be applied daily for 3 months in all females). the females in the second group will be waiting-list control females.

ELIGIBILITY:
Inclusion Criteria:

* systemic sclerosis women (40 females)

Exclusion Criteria:

* obesity
* thoracic diseases
* heart disease
* females with mental diseases

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
cortisol | 12 weeks
  a hormone that is usually represents as a stress hormone

SECONDARY OUTCOMES:
systolic blood pressure | 12 weeks
  it will be measured by sphygmomanometer
diastolic blood pressure | 12 weeks
  it will be measured by sphygmomanometer
pulse rate | 12 weeks
  rate of pulse per minute
respiratory rate | 12 weeks
  rate of respiration per minute
Patient Health Questionnaire | 12 weeks
  it contains eight questions. it will used to assess depression
Hamilton Anxiety Rating Scale | 12 weeks
  a psychological questionnaire used to assess psychological satus
fatigue using visual analogue scale | 12 weeks
  it will be measured using visual analogue scale
Pittsburgh Sleep Quality Index | 12 weeks
  it will measured the sleeping quality of females

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt